CLINICAL TRIAL: NCT01964924
Title: A Single Arm, Phase II Study of Single Agent Trametinib Followed by Trametinib in Combination With GSK2141795 in Patients With Advanced Triple Negative Breast Cancer
Brief Title: Trametinib and Akt Inhibitor GSK2141795 in Treating Patients With Metastatic Triple-Negative Breast Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-01895; NCI-2013-01895 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2013C0069; OSU 13117; 9455 (Other: Ohio State University Comprehensive Cancer Center); 9455 (Other: CTEP); N01CM00070 (NIH); N01CM00100 (NIH); P30CA016058 (NIH); UM1CA186712 (NIH); UM1CA186716 (NIH)
Record Dates: First submitted 2013-10-15; First posted 2013-10-17 (Estimated); Results first posted 2019-09-20 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-08

CONDITIONS: Estrogen Receptor Negative; HER2/Neu Negative; Invasive Breast Carcinoma; Progesterone Receptor Negative; Recurrent Breast Carcinoma; Stage IV Breast Cancer; Triple-Negative Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms | interventions — GSK2141795; trametinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (trametinib, Akt inhibitor GSK2141795) (Experimental): PART 1: Patients receive trametinib PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients who experience disease progression continue to Part 2.
  PART 2: Patients receive trametinib as in Part 1 and also receive Akt inhibitor GSK2141795 PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Akt Inhibitor GSK2141795; Other: Laboratory Biomarker Analysis; Drug: Trametinib

INTERVENTIONS:
Drug: Akt Inhibitor GSK2141795 — Given PO
  Other Names: GSK2141795; Oral Akt Inhibitor GSK2141795
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Trametinib — Given PO
  Other Names: GSK1120212; JTP-74057; MEK Inhibitor GSK1120212; Mekinist

SUMMARY:
This phase II trial studies how well trametinib and v-akt murine thymoma viral oncogene homolog 1 (Akt) inhibitor GSK2141795 work in treating patients with triple-negative breast cancer (breast cancer cells that do not have estrogen receptors, progesterone receptors, or large amounts of human epidermal growth factor receptor 2 [HER2/neu] protein) that has spread to other places in the body. Trametinib and Akt inhibitor GSK2141795 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the anti-tumor activity associated with trametinib monotherapy in patients with triple negative breast cancer (TNBC).

SECONDARY OBJECTIVES:

I. To assess the anti-tumor activity associated with trametinib in combination with AKT inhibitor GSK2141795 after progression on trametinib in patients with metastatic TNBC.

II. To determine the progression-free survival following the initiation of treatment with trametinib monotherapy in patients with metastatic TNBC.

III. To determine the progression-free survival following the initiation of treatment with trametinib in combination with GSK2141795 in patients with metastatic TNBC.

IV. To determine the overall survival following the initiation of treatment with trametinib with GSK214179 in patients with metastatic TNBC.

V. To determine the nature and degree of toxicities associated with trametinib monotherapy and trametinib in combination with GSK2141795 in patients with metastatic TNBC.

VI. To determine the biomarker potential of phosphatase and tensin homolog (PTEN) to predict response to single agent trametinib.

VII. To determine molecular markers of sensitivity and resistance to trametinib monotherapy and trametinib in combination with GSK2141795 in patients with metastatic TNBC.

OUTLINE:

PART 1: Patients receive trametinib orally (PO) once daily (QD) on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients who experience disease progression continue to Part 2.

PART 2: Patients receive trametinib as in Part 1 and also receive Akt inhibitor GSK2141795 PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed metastatic invasive breast cancer that is negative for the estrogen receptor (ER), progesterone receptor (PR) and HER2 by institutional guidelines
* Patients must have measurable disease (Response Evaluation Criteria in Solid Tumors version 1.1 [RECIST 1.1])
* Patients must have had exposure to at least 1 and no more than 3 prior chemotherapy regimens for the treatment of metastatic breast cancer
* Patients must consent to both a pretreatment and a post-treatment mandatory research biopsy prior to enrolling on trial, and therefore, must have tissue (excluding bone or brain) that is amenable to biopsy
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1
* Life expectancy of greater than 3 months
* Able to swallow and retain orally administered medication and does not have any clinically significant gastrointestinal abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach or bowels
* All prior treatment-related toxicities must be Common Terminology Criteria for Adverse Events version 4 (CTCAE v4) grade =< 1 (except alopecia) at the time of enrollment
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 75,000/mcL
* Total bilirubin =< 1.5 × institutional upper limit of normal
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 × institutional upper limit of normal
* Left ventricular ejection fraction (LVEF) >= institutional lower limit of normal by echocardiogram (ECHO) or multiple gated acquisition scan (MUGA)
* Serum creatinine =< 1.5 mg/dL OR calculated creatinine clearance (Cockcroft-Gault formula) >= 50 mL/min OR 24-hour urine creatinine clearance >= 50 mL/min
* Patients must have controlled blood pressure with a systolic blood pressure < 140 mmHg and diastolic < 90 mmHg; anti-hypertensive medications are permitted
* Patients must be at least 4 weeks from last radiation dose; patients must be at least 4 weeks from last chemotherapy, targeted therapy, or biologic therapy (exception allowed for a 2 week washout for patients who were on chemotherapy at less than a standard of care dose, as long as all other eligibility criteria are met); patients must be at least 4 weeks from last surgical procedure and recovered from all post-operative complications
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of trametinib monotherapy or in combination with GSK2141795 administration
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* History of another malignancy

  * Exception: patients who have been disease-free for 3 years, or patients with a history of completely resected non-melanoma skin cancer and/or patients with indolent secondary malignancies, are eligible
* History of interstitial lung disease or pneumonitis
* History of type I diabetes mellitus; if a patient has type II diabetes, they must have a hemoglobin (hemoglobin A1C) =< 8%; patients with a screening fasting glucose > 120 mg/dL will be excluded
* Uncontrolled hypothyroidism; patients must have a normal thyroid-stimulating hormone (TSH) per institutional standards at baseline
* Patients who are receiving any other investigational agents
* Individuals with symptomatic or progressive brain metastases are ineligible; subjects with treated brain metastases are eligible if they have no radiographic or other signs of progression in the brain for >= 3 weeks after completion of local therapy; any corticosteroid use for brain metastases must have been discontinued without the subsequent appearance of symptoms for >= 3 weeks prior to study enrollment
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to trametinib monotherapy or trametinib in combination with GSK2141795
* Current use of a prohibited medication; the following medications or non-drug therapies are prohibited:

  * Other anti-cancer therapy while on study treatment (megestrol if used as an appetite stimulant is allowed)
  * The concurrent use of all herbal supplements is prohibited during the study (including, but not limited to, St. John's wort, kava, ephedra [ma huang], gingko biloba, yohimbe, saw palmetto, or ginseng)
  * Patients receiving strong inhibitors or inducers of cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) are ineligible
* History or current evidence/risk of retinal vein occlusion (RVO) or central serous retinopathy (CSR) or predisposing factors to RVO or CSR (e.g., uncontrolled glaucoma or ocular hypertension, uncontrolled hypertension, history of hyperviscosity or hypercoagulability syndromes; visible retinal pathology as assessed by ophthalmic exam that is considered a risk factor for RVO or CSR such as evidence of new optic disc cupping, evidence of new visual field defects, and intraocular pressure > 21 mm Hg
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study, breastfeeding should be discontinued if the mother is treated with trametinib monotherapy or trametinib in combination with GSK2141795
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2013-10-02 (Actual); Primary Completion 2017-01-20 (Actual); Study Completion 2018-04-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bhuvaneswari Ramaswamy, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (8):
- United States (8):
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Moffitt Cancer Center, Tampa, Florida
  - Roswell Park Cancer Institute, Buffalo, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients on Part 1: trametinib monotherapy until progression and then will continue on to Part 2: trametinib combined with GSK2141795.
Groups:
- Treatment (Trametinib, Akt Inhibitor GSK2141795) PART 1:: PART 1: Patients receive trametinib PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients who experience disease progression in Part 1 continue to Part 2.
- Treatment (Trametinib, Akt Inhibitor GSK2141795) PART 2:: PART 2: Patients who experience disease progression in Part 1 continue to Part 2. Patients receive trametinib and also receive Akt inhibitor GSK2141795 PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Akt Inhibitor GSK2141795: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Trametinib: Given PO
Period: Trametinib Monotherapy
Arm/Group | Treatment (Trametinib, Akt Inhibitor GSK2141795) PART 1: | Treatment (Trametinib, Akt Inhibitor GSK2141795) PART 2:
Started | 37 | 0
Completed | 18 | 0
Not Completed | 19 | 0
Not completed — Progression | 19 | 0
Period: Trametinib + GSK2141
Arm/Group | Treatment (Trametinib, Akt Inhibitor GSK2141795) PART 1: | Treatment (Trametinib, Akt Inhibitor GSK2141795) PART 2:
Started (Participants who completed Part 1 were not eligible for Part 2) | 0 | 19 (Progressed in Part 1 and therefore initiated combination treatment in Part 2)
Completed | 0 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment (Trametinib, Akt Inhibitor GSK2141795): PART 1: Patients receive trametinib PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients who experience disease progression continue to Part 2.
  PART 2: Patients receive trametinib as in Part 1 and also receive Akt inhibitor GSK2141795 PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Akt Inhibitor GSK2141795: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Trametinib: Given PO
Arm/Group | Treatment (Trametinib, Akt Inhibitor GSK2141795)
Number analyzed (Participants) | 37
Age, Continuous [Median (Full Range); unit: years] | 57 [35 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 37
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 31
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 37

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR), Defined as the Proportion of Patients Who Have Had a Partial Response (PR) or Complete Response (CR) (RECIST 1.1 Based) Within the First 6 Months After Initiation of Therapy With Trametinib
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Trametinib, Akt Inhibitor GSK2141795)
Number analyzed (Participants) | 37
Participants | 2

2. Secondary Outcome: Clinical Benefit Rate (CBR = CR+PR+Stable Disease [SD])
Description: The clinical benefit rate (CR+PR+SD) will be reported for patients after Part 1 and after Part 2.
Time Frame: Up to 52 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Treatment (Trametinib, Akt Inhibitor GSK2141795) PART 1:: PART 1: Patients receive trametinib PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients who experience disease progression continue to Part 2.
- Treatment (Trametinib, Akt Inhibitor GSK2141795) PART 2:: PART 2: Patients receive trametinib as in Part 1 and also receive Akt inhibitor GSK2141795 PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Akt Inhibitor GSK2141795: Given PO
  Laboratory Biomarker Analysis: Correlative studies
  Trametinib: Given PO
Arm/Group | Treatment (Trametinib, Akt Inhibitor GSK2141795) PART 1: | Treatment (Trametinib, Akt Inhibitor GSK2141795) PART 2:
Number analyzed (Participants) | 37 | 19
Participants | 8 | 6

3. Secondary Outcome: Duration of Objective Response
Description: Summary statistics of duration of response for patients with objective response
Time Frame: up to 52 weeks
Measure: Mean (Standard Deviation); unit: days of response
Arm/Group | Treatment (Trametinib, Akt Inhibitor GSK2141795) PART 1: | Treatment (Trametinib, Akt Inhibitor GSK2141795) PART 2:
Number analyzed (Participants) | 8 | 6
days of response | 162.75 (149.26) | 87.00 (62.86)

4. Secondary Outcome: Incidence of Adverse Events That Are Classified as Either Possibly, Probably, or Definitely Related to Study Treatment
Description: Incidence of adverse events for patients that are classified as either possibly, probably, or definitely related to study treatment graded by National Cancer Institute (NCI) CTCAE v4.0
Time Frame: Up to 52 weeks
Measure: Number; unit: number of adverse events
Groups:
- Treatment (Trametinib, Akt Inhibitor GSK2141795) PART 2:: PART 2: Patients receive trametinib as in Part 1 and also receive Akt inhibitor GSK2141795 PO QD on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Arm/Group | Treatment (Trametinib, Akt Inhibitor GSK2141795) PART 1: | Treatment (Trametinib, Akt Inhibitor GSK2141795) PART 2:
Number analyzed (Participants) | 37 | 19
number of adverse events | 227 | 204

5. Secondary Outcome: Incidence of Severe (Grade 3+) Adverse Events or Toxicities Graded Per NCI CTCAE Version 4.0
Description: NCI CommonTerminology Criteria for Adverse Events (CTCAE) version 4.0 was utilized for grading incidence of toxicities (grade 3+).
Time Frame: Up to 52 weeks
Measure: Number; unit: number of adverse events
Arm/Group | Treatment (Trametinib, Akt Inhibitor GSK2141795) PART 1: | Treatment (Trametinib, Akt Inhibitor GSK2141795) PART 2:
Number analyzed (Participants) | 37 | 19
number of adverse events | 68 | 29

6. Secondary Outcome: Overall Survival
Description: The Kaplan-Meier method will be used to estimate overall survival distribution.
Time Frame: Start date of the treatment to the date of the event (i.e., death) or the date of last follow-up to evaluate that event, assessed up to 52 weeks
Population: overall survival analyzed for all patients regardless of (part 1 only) or (part 1 and 2) participation
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Treatment (Trametinib, Akt Inhibitor GSK2141795)
Number analyzed (Participants) | 37
weeks | 43.143 [33.0 to 99.286]

7. Secondary Outcome: Progression-free Survival
Description: The Kaplan-Meier method will be used to estimate progression-free survival distribution.
Time Frame: The duration of time from start of treatment to time of progression or death, whichever comes first, assessed up to 52 weeks
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Treatment (Trametinib, Akt Inhibitor GSK2141795) PART 1: | Treatment (Trametinib, Akt Inhibitor GSK2141795) PART 2:
Number analyzed (Participants) | 37 | 19
weeks | 7.71 [4.43 to 8.29] | 7.86 [5.86 to 13.86]

8. Secondary Outcome: Proportion of Patients Who go Off Treatment Due to Adverse Reactions
Description: The proportion of patients who go off treatment due to adverse reactions or even those who refuse further treatment for lesser toxicities that inhibit their willingness to continue participation on the trial was captured. These tolerability measures were assessed within each of the treatment parts independently. All patients who have received at least one dose of any of the therapeutic agents was evaluable for toxicity and tolerability.
Time Frame: Up to 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Trametinib, Akt Inhibitor GSK2141795) | Treatment (Trametinib, Akt Inhibitor GSK2141795) PART 2:
Number analyzed (Participants) | 37 | 19
Participants | 4 | 0

9. Secondary Outcome: Proportion of Patients Who Refuse Further Treatment for Lesser Toxicities That Inhibit Their Willingness to Continue Participation on the Trial
Time Frame: Up to 52 weeks
Population: The proportion of patients who refuse further treatment for lesser toxicities that inhibit their willingness to continue participation on the trial was in Part I
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Trametinib, Akt Inhibitor GSK2141795) | Treatment (Trametinib, Akt Inhibitor GSK2141795) PART 2:
Number analyzed (Participants) | 37 | 0
Participants | 2 | 0

10. Secondary Outcome: Tolerability of the Regimen Defined as the Number of Patients Who Required Dose Modifications and/or Dose Delays
Time Frame: Up to 52 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Trametinib, Akt Inhibitor GSK2141795) | Treatment (Trametinib, Akt Inhibitor GSK2141795) PART 2:
Number analyzed (Participants) | 37 | 19
Participants | 35 | 0

11. Other Pre Specified Outcome: Predictive Value of PTEN and Other Biomarkers on Patient Outcome (Survival, ORR, and CBR)
Time Frame: At time of disease progression, assessed up to 52 weeks
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Protein Intensity Fold-change Ratios Assessed by Reverse Phase Protein Assay Intensity Values
Description: Ratios between tumors sampled prior to initiating trametinib single agent treatment and at time of progression (TOP) on either single agent trametinib or the combination (TOP/pre-treat ratio), will be calculated. These ratios will be median-centered and clustered using Cluster 2.0 software. Student's t-test for differences between average protein intensity ratios at these intervals will be calculated using Microsoft Excel by grouping all the ratios for individual clusters.
Time Frame: Up to 52 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 1 year patients will be evaluated for toxicities from the time of their first treatment until they are off study.
Description: Adverse Event grading was done using NCI CTCAE version 4.0
Arm/Group | Treatment (Trametinib, Akt Inhibitor GSK2141795) PART 1: | Treatment (Trametinib, Akt Inhibitor GSK2141795) PART 2:
All-Cause Mortality (participants affected / at risk) | 13/37 | 12/19
Serious Adverse Events (participants affected / at risk) | 30/37 | 15/19
Other Adverse Events (participants affected / at risk) | 37/37 | 19/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Trametinib, Akt Inhibitor GSK2141795) PART 1: (N=37) | Treatment (Trametinib, Akt Inhibitor GSK2141795) PART 2: (N=19)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Death NOS (General disorders) | 1 (1) | 4 (4)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Edema face (General disorders) | 1 (1) | 0 (0)
Edema limbs (General disorders) | 1 (1) | 0 (0)
Enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Fever (General disorders) | 1 (1) | 1 (1)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglossal nerve disorder (Nervous system disorders) | 1 (1) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 8 (8) | 3 (3)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 2 (2) | 0 (0)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Trametinib, Akt Inhibitor GSK2141795) PART 1: (N=37) | Treatment (Trametinib, Akt Inhibitor GSK2141795) PART 2: (N=19)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 0 (0)
Alanine aminotransferase increased (Investigations) | 7 (7) | 2 (2)
Alkaline phosphatase increased (Investigations) | 6 (6) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 7 (7) | 8 (8)
Anorexia (Metabolism and nutrition disorders) | 5 (5) | 2 (2)
Anxiety (Psychiatric disorders) | 4 (4) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 13 (13) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4)
Blurred vision (Eye disorders) | 1 (1) | 2 (2)
Breast pain (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 5 (5) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Creatinine increased (Investigations) | 4 (4) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 5 (5)
Depression (Psychiatric disorders) | 4 (4) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 11 (11) | 16 (16)
Dizziness (Nervous system disorders) | 3 (3) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 4 (4) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 5 (5) | 4 (4)
Dysgeusia (Nervous system disorders) | 0 (0) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 5 (5)
Dysphasia (Nervous system disorders) | 0 (0) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 (9) | 8 (8)
Edema face (General disorders) | 4 (4) | 1 (1)
Edema limbs (General disorders) | 11 (11) | 4 (4)
Edema trunk (General disorders) | 2 (2) | 0 (0)
Ejection fraction decreased (Investigations) | 0 (0) | 1 (1)
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 (0) | 2 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3)
Esophageal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Facial pain (General disorders) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Fatigue (General disorders) | 11 (11) | 6 (6)
Fever (General disorders) | 3 (3) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Flu like symptoms (General disorders) | 2 (2) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 2 (2) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2)
Headache (Nervous system disorders) | 4 (4) | 0 (0)
Heart failure (Cardiac disorders) | 1 (1) | 1 (1)
Hematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 7 (7) | 6 (8)
Hypertension (Vascular disorders) | 5 (5) | 7 (9)
Hyperthyroidism (Endocrine disorders) | 2 (2) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 9 (9) | 7 (8)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (3) | 4 (5)
Hypoglycemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 3 (3) | 2 (6)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 3 (3) | 1 (3)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 1 (1) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
INR increased (Investigations) | 0 (0) | 1 (1)
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) | 3 (4)
Insomnia (Psychiatric disorders) | 2 (2) | 2 (2)
Investigations - Other, specify (Investigations) | 0 (0) | 2 (3)
Left ventricular systolic dysfunction (Cardiac disorders) | 1 (1) | 1 (1)
Localized edema (General disorders) | 1 (1) | 1 (1)
Lymphedema (Vascular disorders) | 5 (5) | 2 (2)
Lymphocyte count decreased (Investigations) | 6 (6) | 4 (4)
Movements involuntary (Nervous system disorders) | 0 (0) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 4 (4) | 12 (13)
Nail ridging (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 12 (12) | 5 (6)
Neck edema (General disorders) | 2 (2) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neoplasms benign, malignant and unspecified (incl cysts and polyps-Other (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 2 (2)
Neutrophil count decreased (Investigations) | 1 (1) | 2 (3)
Non-cardiac chest pain (General disorders) | 2 (2) | 3 (3)
Pain (General disorders) | 4 (4) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 (4) | 2 (2)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Paronychia (Infections and infestations) | 1 (1) | 2 (2)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 5 (5) | 4 (4)
Platelet count decreased (Investigations) | 7 (7) | 3 (3)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
Presyncope (Nervous system disorders) | 0 (0) | 1 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 6 (6) | 3 (5)
Rash acneiform (Skin and subcutaneous tissue disorders) | 10 (10) | 3 (5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 (6) | 3 (3)
Sinus tachycardia (Cardiac disorders) | 3 (3) | 0 (0)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 4 (4) | 3 (3)
Skin infection (Infections and infestations) | 2 (2) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Thromboembolic event (Vascular disorders) | 0 (0) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 2 (2) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 6 (6) | 3 (3)
Weight gain (Investigations) | 3 (3) | 1 (1)
Weight loss (Investigations) | 1 (1) | 3 (4)
White blood cell decreased (Investigations) | 5 (5) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-30): https://cdn.clinicaltrials.gov/large-docs/24/NCT01964924/Prot_SAP_000.pdf